CLINICAL TRIAL: NCT05918068
Title: Evaluation of the Role of Pyridoxine Adjuvant Therapy on the Blood Glucose Level in Type 2 Diabetic Patients
Brief Title: Pyridoxine Effect on the Blood Glucose Level in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Rasheed University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AR200108
Record Dates: First submitted 2023-05-30; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Vitamin B 6; Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): Newly diagnosed patients with T2DM, treated with non-pharmacological therapy (lifestyle modification).
  Interventions: Other: non-pharmacological therapy
- Metformin only group (Active Comparator): T2DM patients treated with metformin 500 mg/day in addition to non-pharmacological therapy (lifestyle modification)
  Interventions: Drug: Metformin 500 mg/day; Other: non-pharmacological therapy
- Combination group (Experimental): T2DM patients treated with metformin 500 mg/day plus vitamin B6 300 mg/day in addition to non-pharmacological therapy (lifestyle modification)
  Interventions: Drug: Metformin 500 mg/day; Combination Product: Metformin 500 mg/day plus vitamin B6 300 mg/day; Other: non-pharmacological therapy

INTERVENTIONS:
Drug: Metformin 500 mg/day — Metformin 500 mg/day in addition to non-pharmacological therapy
  Other Names: Metformin group
  Arms: Combination group; Metformin only group
Combination Product: Metformin 500 mg/day plus vitamin B6 300 mg/day — Metformin 500 mg/day plus vitamin B6 300 mg/day in addition to non-pharmacological therapy
  Other Names: Combination group
  Arms: Combination group
Other: non-pharmacological therapy — non-pharmacological therapy (healthy lifestyle modifications)
  Other Names: control group

SUMMARY:
Pyridoxal-5-phosphate (P.L.P.), the biologically active form of vitamin B6, is a coenzyme in 150 enzymatic reactions, including amino acid, carbohydrate, and lipid metabolism. Neurotransmitter production and breakdown depend on it. Additionally, it functions as an antioxidant by suppressing reactive oxygen species and mitigating the development of advanced glycation end products. Humans recycle P.L.P. from dietary B6 vitamins, and this molecule has been related to various clinically relevant diseases. Pyridoxine as an additional therapy for type 2 diabetes will be examined in this study.

DETAILED DESCRIPTION:
Numerous organs might suffer long-term harm, malfunction, and failure as a result of type 2 diabetes. While the illness may initially cause weight loss, frequent urination, thirst, and hazy vision, the long-term repercussions may include the gradual onset of specific issues such as cardiovascular disease (CVD), retinopathy, which may culminate in blindness, and renal disease. The risk of foot ulcers, Charcot joints, and symptoms of autonomic dysfunction, such as sexual dysfunction, is associated with renal failure and/or neuropathy. Diabetes and vitamin B6 have both been linked. It is not apparent, therefore, whether diabetes is a consequence of low P.L.P. levels, a cause, or both. According to some study, diabetes may develop as a consequence of low P.L.P. levels, however other studies suggest that diabetes decreases P.L.P. levels. Although the physiological and molecular pathways behind these beneficial effects on diabetic pathology and related repercussions are not completely understood, multiple investigations have demonstrated that B6 therapy has good effects. There are numerous ways that pyridoxal 5-phosphate deficiency affects diabetes. As an essential element for numerous enzymes that contribute to this process, pyridoxal-5-phosphate can, for example, influence the route that converts tryptophan into niacin. It has been proven that the metabolites produced when this pathway is damaged lessen the bioactivity of insulin and cause insulin resistance, a T2D symptom . Pyridoxal-5-phosphate may influence insulin resistance via modulating the expression of adipogenesis-related genes. The degradation of co-enzyme-dependent enzymes like (C.B.S.) and (C.G.L.), which rely on pyridoxal-5-phosphate, may also promote insulin resistance via elevating homocysteine levels .

This research intends to examine the impact of pyridoxine adjuvant treatment on the blood glucose level in type 2 diabetes patients.

This is a randomized controlled open-label interventional study. T2DM patients who receive either (metformin with pyridoxine) or (metformin only) daily and T2DM patients treated with non-pharmacological therapy (lifestyle modification) will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes mellitus newly diagnosed patient with age (Above 30) years.
* HbA1c less than or equal to 7.5%.

Exclusion Criteria:

* Type 1 Diabetes mellitus.
* Concomitant chronic diseases (Rheumatoid arthritis, anemia, asthma, endocrine disorders, renal failure, alcoholics, and patient on anti-T.B. or anti-epileptics).
* Females should be neither pregnant nor on oral contraceptive drugs.
* Not taking any vitamin or mineral supplementation.
* Should have no history of recent acute infection (within the previous two weeks).

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Fasting plasma glucose (FPG). | Change from baseline, to one month
  A fasting plasma glucose test, also known as a fasting glucose test (FGT), is a test that can be used to help diagnose diabetes or pre-diabetes.The expected values for normal fasting blood glucose concentration are between 70 mg/dL (3.9 mmol/L) and 100 mg/dL (5.6 mmol/L). When fasting blood glucose is between 100 to 125 mg/dL (5.6 to 6.9 mmol/L), changes in lifestyle and monitoring glycemia are recommended
Glycated Hemoglobin (HbAlc) | Change from baseline, to one month
  A normal A1C level is below 5.7%, a level of 5.7% to 6.4% indicates prediabetes and a level of 6.5% or more indicates diabetes.

SECONDARY OUTCOMES:
Vitamin B6 | Change from baseline, to one month
  The reference range for pyridoxal phosphate (PLP), the biologically active form of vitamin B6, is 5-50 µg/L.
Fasting plasma insulin (F.P.I.). | Change from baseline, to one month
  The insulin fasting blood test is chiefly used to test insulin levels and diagnose diabetes and insulin resistance.
Insulin resistance (HOMA-IR). | Change from baseline, to one month
  Less than 1.0 means you are insulin-sensitive which is optimal. Above 1.9 indicates early insulin resistance. Above 2.9 indicates significant insulin resistance.
Indoleamine 2,3 dioxygenase (IDO) | Change from baseline, to one month
  Has the potential role of indoleamine 2,3 dioxygenase (IDO) as a predictive and therapeutic target for diabetes treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Maysan Centre for Diabetes and Endocrinology, Maysan Governorate, Iraq

REFERENCES:
- [Background] Mascolo E, Verni F. Vitamin B6 and Diabetes: Relationship and Molecular Mechanisms. Int J Mol Sci. 2020 May 23;21(10):3669. doi: 10.3390/ijms21103669. PMID 32456137
- [Background] Merigliano C, Mascolo E, Burla R, Saggio I, Verni F. The Relationship Between Vitamin B6, Diabetes and Cancer. Front Genet. 2018 Sep 13;9:388. doi: 10.3389/fgene.2018.00388. eCollection 2018. PMID 30271425
- [Background] Petersmann A, Muller-Wieland D, Muller UA, Landgraf R, Nauck M, Freckmann G, Heinemann L, Schleicher E. Definition, Classification and Diagnosis of Diabetes Mellitus. Exp Clin Endocrinol Diabetes. 2019 Dec;127(S 01):S1-S7. doi: 10.1055/a-1018-9078. Epub 2019 Dec 20. No abstract available. PMID 31860923